CLINICAL TRIAL: NCT00119847
Title: Electrophysiological Effects of Late PCI (OAT-EP)
Brief Title: Electrophysiological Effects of Late PCI After MI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Eric Rashba, Associate Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 221; R01HL072906 (NIH)
Record Dates: First submitted 2005-07-06; First posted 2005-07-14 (Estimated); Results first posted 2018-08-23 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Myocardial Infarction; Coronary Disease; Arrhythmia; Ventricular Fibrillation
Keywords: Stents, myocardial infarction
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Myocardial Infarction; Coronary Disease; Arrhythmias, Cardiac; Ventricular Fibrillation | interventions — Angioplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PCI+MED (Experimental): Percutaneous Coronary Intervention (PCI) with angioplasty and stenting of the infarct-related artery and optimal medical therapy
  Interventions: Procedure: PCI; Drug: Optimal Medical Therapy
- MED (Experimental): Optimal medical therapy alone
  Interventions: Drug: Optimal Medical Therapy

INTERVENTIONS:
Procedure: PCI
  Other Names: Angioplasty and stenting of the infarct-related artery
  Arms: PCI+MED
Drug: Optimal Medical Therapy — Guideline-directed drug therapies after MI

SUMMARY:
The purpose of this study is to determine if opening blocked arteries with heart balloons and stents prevents heart rhythm problems in individuals 3 to 28 days after a heart attack.

DETAILED DESCRIPTION:
BACKGROUND:

There is now unequivocal evidence that early coronary reperfusion using either thrombolytics or primary angioplasty results in a long-term mortality reduction among individuals who have had a heart attack. The benefit of early reperfusion (less than 6 hours after the heart attack) was initially attributed to myocardial salvage and the resultant preservation of left ventricular function. However, it is now known that the survival benefit associated with thrombolytic therapy is not consistently associated with a major improvement in left ventricular ejection fraction (LVEF). These observations led to the formulation of the "late open artery hypothesis," which suggests that clinical outcomes can potentially be improved by late reperfusion after a heart attack. Observational clinical studies have suggested that late patency of the infarct-related artery (IRA) after thrombolysis is associated with a survival benefit that is independent of LVEF and therefore cannot be solely explained by salvage of myocardium. Definitive proof of the late open artery hypothesis is currently lacking, however, because previous studies that have evaluated late percutaneous transluminal coronary angioplasty (PTCA) of occluded IRAs after a heart attack have produced conflicting results.

These findings led to the organization of the Occluded Artery Trial (OAT), an international, NHLBI-funded, randomized trial of 2,200 participants. OAT is testing the hypothesis that mechanical reperfusion of an occluded IRA with PTCA and percutaneous coronary intervention (PCI) 3 to 28 days after a heart attack in high-risk individuals will reduce mortality, recurrent heart attacks, and hospitalization for class IV congestive heart failure. Enhancement of electrical stability is one of the major mechanisms that has been proposed to explain the association of an open IRA with an improved prognosis independent of myocardial salvage.

DESIGN NARRATIVE:

This study is an ancillary study of OAT. It will characterize the effects of late PCI of occluded IRAs on the most important and clinically relevant noninvasive markers of vulnerability to malignant ventricular arrhythmias: heart rate variability, T wave variability, and signal-averaged electrocardiography. These analyses will be performed in 300 participants at baseline, 30 days, and 1 year following a heart attack in order to determine the effects of late PCI on the autonomic nervous system, ventricular repolarization, and ventricular conduction abnormalities.

ELIGIBILITY:
Inclusion Criteria:

* Has experienced a heart attack 3 to 28 days prior to study entry
* Persistently occluded IRA defined as either: 1) Thrombolysis in Myocardial Infarction (TIMI) 0, with no flow beyond the site of occlusion; or 2) TIMI 1, with penetration of dye beyond the site of occlusion without dye reaching the distal vessel
* LVEF less than 50% or proximal occlusion in a large vessel
* Normal sinus rhythm
* QRS duration less than 120 ms
* Able to return for follow-up assessment of arrhythmia markers one month and one year after study entry

Exclusion Criteria:

* Has a clinical indication for revascularization (post-heart attack angina at rest; significant inducible ischemia; or significant left main or triple vessel disease requiring PTCA or CABG)
* Current serious illness or condition that limits 3-year survival
* Severe valvular disease
* Chronic total occlusion
* New York Heart Association Class III-IV congestive heart failure
* Prior left ventricular aneurysm in the recent heart attack location
* Is a poor candidate for PTCA/stent on the basis of angiographic or clinical criteria
* Cannot medically survive anticoagulation during PTCA/stent or antiplatelet therapy after stent
* Pregnant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2002-09 (Actual); Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric J. Rashba, MD, Study Chair — Stony Brook University Medical Center
Locations (1):
- Stony Brook University Medical Center, Stony Brook, New York, United States

REFERENCES:
- [Background] Rashba EJ. Assessment of ventricular repolarization abnormalities in congenital long QT syndrome. J Cardiovasc Electrophysiol. 2004 May;15(5):557-9. doi: 10.1046/j.1540-8167.2004.04022.x. No abstract available. PMID 15149425
- [Background] Rashba EJ. Should T-wave alternans testing be used to risk stratify candidates for prophylactic implantable cardioverter-defibrillator therapy? Heart Rhythm. 2005 Mar;2(3):242-4. doi: 10.1016/j.hrthm.2004.12.015. No abstract available. PMID 15851311
- [Result] Rashba EJ, Lamas GA, Couderc JP, Hollist SM, Dzavik V, Ruzyllo W, Fridrich V, Buller CE, Forman SA, Kufera JA, Carvalho AC, Hochman JS; OAT-EP Investigators. Electrophysiological effects of late percutaneous coronary intervention for infarct-related coronary artery occlusion: the Occluded Artery Trial-Electrophysiological Mechanisms (OAT-EP). Circulation. 2009 Feb 17;119(6):779-87. doi: 10.1161/CIRCULATIONAHA.108.808626. Epub 2009 Feb 2. PMID 19188505

RESULTS

PARTICIPANT FLOW:
Groups:
- PCI+Optimal Medical Therapy: PCI with angioplasty and stenting of the infarct-related artery and optimal medical therapy
  Optimal Medical Therapy: Guideline-directed drug therapies after MI
- Optimal Medical Therapy: Optimal medical therapy alone
  Optimal Medical Therapy: Guideline-directed drug therapies after MI
Period: Overall Study
Arm/Group | PCI+Optimal Medical Therapy | Optimal Medical Therapy
Started | 149 | 151
Completed | 118 | 119
Not Completed | 31 | 32

BASELINE CHARACTERISTICS:
Groups:
- PCI+Optimal Medical Therapy: PCI with angioplasty and stenting of the infarct-related artery and optimal medical therapy
  PCI
  Optimal Medical Therapy: Guideline-directed drug therapies after MI
- Total: Total of all reporting groups
Arm/Group | PCI+Optimal Medical Therapy | Optimal Medical Therapy | Total
Number analyzed (Participants) | 149 | 151 | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (10.5) | 57.6 (10.5) | 57.4 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 24 | 62
  Male | 111 | 127 | 238
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 115 | 117 | 232
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 31 | 30 | 61

OUTCOME MEASURES:

1. Primary Outcome: Short-termed Fractal Scaling Exponent (Alpha 1)
Description: Nonlinear measurement of heart rate variability, change between baseline and 1 year is the primary outcome.
Time Frame: Baseline, one year
Measure: Mean (Standard Deviation); unit: unit-less
Arm/Group | PCI+Optimal Medical Therapy | Optimal Medical Therapy
Number analyzed (Participants) | 118 | 119
unit-less | 0.01 (0.34) | -0.03 (0.32)
Statistical Analysis 1: Comparison: PCI+Optimal Medical Therapy vs Optimal Medical Therapy; The planned sample size of 300 subjects was chosen to provide 80% power to detect a clinically relevant difference of 0.1 in the change in α1 from baseline to 1 year between the 2 treatment groups on the basis of data from prior studies that indicated that baseline levels of α1 would be 1.0 with a common SD of 0.2; Test type: Superiority; p = 0.34, t-test, 2 sided — p<0.05 required for statistical significance; Mean Difference (Net) = -0.04, 95% CI 2-sided [-0.12 to 0.04]

2. Secondary Outcome: T-wave Variability
Description: Variability in T wave morphology, change between baseline and one year
Time Frame: Baseline and one year
Measure: Mean (Standard Deviation); unit: Microvolts
Arm/Group | PCI+Optimal Medical Therapy | Optimal Medical Therapy
Number analyzed (Participants) | 104 | 103
Microvolts | -6.3 (25.1) | -3.4 (31.0)
Statistical Analysis 1: Comparison: PCI+Optimal Medical Therapy vs Optimal Medical Therapy; Test type: Superiority; p = 0.45, t-test, 2 sided — p<0.01 required for statistical significance; Mean Difference (Net) = 3.0, 95% CI 2-sided [-4.8 to 10.7]

3. Secondary Outcome: Filtered QRS Duration
Description: Signal-averaged ECG
Time Frame: Baseline and one year
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | PCI+Optimal Medical Therapy | Optimal Medical Therapy
Number analyzed (Participants) | 90 | 81
Milliseconds | 1.5 (12.4) | 3.7 (11.8)
Statistical Analysis 1: Comparison: PCI+Optimal Medical Therapy vs Optimal Medical Therapy; Test type: Superiority; p = 0.23, t-test, 2 sided — p<0.01 required for statistical significance; Mean Difference (Net) = 2.2, 95% CI 2-sided [-1.4 to 5.9]

ADVERSE EVENTS:
Arm/Group | PCI+Optimal Medical Therapy | Optimal Medical Therapy
Serious Adverse Events (participants affected / at risk) | 0/149 | 0/151
Other Adverse Events (participants affected / at risk) | 0/149 | 0/151

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No